CLINICAL TRIAL: NCT00327197
Title: A Study to Assess Disease Pathology and Key Therapeutic Targets in Severe Asthma
Brief Title: Assessment Of Disease Pathology And Key Therapeutic Targets In Severe Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was truncated due to the long period of enrollment and the collection of a sufficient amount of data that allowed the scientific objectives to be met
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RES100769
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: bronchoscopy; Sputum induction; Prednisolone; Asthma; biomarkers
MeSH Terms: conditions — Asthma | interventions — Prednisolone; Bronchoscopy

ARMS (4):
- Intermittent mild steroid-naïve asthmatic group (Experimental): Asymptomatic subjects receiving only beta-agonist inhaler with predicted FEV1 >=80% and normal peak expiratory flow between attacks will be included.
  Interventions: Drug: Prednisolone; Procedure: Bronchoscopy
- Mild to moderate persistent asthmatic group (Experimental): Subjects with mild to moderate persistent asthma on low to moderate dose of inhaled corticosteroid (200-500 microgram fluticasone propionate daily or equivalent), an FEV1 >= 80% predicted (post-bronchodilator), and less than 20% variability in peak expiratory flow.
  Interventions: Drug: Prednisolone; Procedure: Bronchoscopy
- Severe asthma group (Experimental): Subjects with severe persistent asthma. They will be on either: high inhaled corticosteroid (CS >=1000 microgram fluticasone daily or equivalent) or on high dose inhaled CS plus oral CS (no more than 20 milligrams predisolone a day). The subjects should have at least one ( if on oral steroids) or two (if only on inhaled steroids) of the following: 1) FEV1<80% and FEV1/FVC ratio <70% 2) more than 25% variability in peak expiratory flow 3) daily symptoms ± nocturnal symptoms 4) severe exacerbations of >= twice a year in at least one of the last two years.
  Interventions: Drug: Prednisolone; Procedure: Bronchoscopy
- Healthy subjects group (Placebo Comparator): Non-asthmatic and non-smokers with FEV1 > 85% predicted, on no regular medication.
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Drug: Prednisolone — Subjects will be administered oral prednisolone at a dose of 0.5 mg/kg, up to a maximum of 40 mg per day for 14 days.
  Arms: Intermittent mild steroid-naïve asthmatic group; Mild to moderate persistent asthmatic group; Severe asthma group
Procedure: Bronchoscopy — All subjects will undergo bronchoscopy assessments which will involve insertion of a standard bronchoscope.

SUMMARY:
To evaluate and compare the expression and change in expression of key severe asthma targets at baseline in mile to moderate asthmatics vs. severe asthmatic subjects.

To evaluate and compare the airway pathology at baseline and changes in airway pathology in relation to asthma severity.

ELIGIBILITY:
Inclusion criteria:

* History of asthma with exclusion of other significant pulmonary disease.
* Body Mass Index between 19-31 kg.m-2.
* Subjects will be assigned to group 1(mild to moderate) or Group 2 (severe asthmatics) depending on their Lung Function test results.

Exclusion criteria:

* As a result of medical interview, physical examination or screening investigation the physician responsible considers the subject unfit for the study.
* History of drug or other allergy, which, in the opinion of the responsible physician, contra-indicates their participation.
* Subject is female who is pregnant or lactating.
* Currently or planning to take during the study regular medication (including over-the-counter) except for medication allowed in inclusion criteria.
* Having participated within 30 days or 5 half-lives, whichever is longer of the first dose in a study using new molecular entity, or the first dose in any other study investigating drugs or having participated within one month of the first dose in a study with invasive procedures.
* History or current evidence of an upper or lower respiratory infection or symptoms (including common cold) within 2 weeks of baseline assessments.
* History of abnormal bruising or bleeding.
* History of alcohol or drug abuse.
* Doing night-shift work within at least 5 days prior to dosing until completion of the study.
* Anticoagulants except low dose of Aspirin (80 mg per day) (for bronchoscopy).
* Beta blockers except for low dose Atenolol (25 mg/day) or Metoprolol (50 mg/day) (for bronchoscopy).
* Use of Cytochrome P450 inhibitors.
* History of hypersensitivity to any of the following medications: Lidocaine, Fentanyl, Versed, Demerol, Midazolam, Epinephrine, Flumazenil and Naloxone.
* History of hypersensitivity to bronchodilator (such as Albuterol).

In addition, the following additional exclusion criteria must apply to mild to moderate persistent asthmatics on regular inhaled steroids:

* Changed asthma medication within the 4 weeks prior to screening.
* Has had an asthma exacerbation in the previous month.
* Known sensitivity or allergy to prednisolone.
* Current use or use within the previous 3 months of oral corticosteroids.
* Current use of Methotrexate, cyclosporine and PDE inhibitors
* History of tuberculosis, diabetes mellitus, osteoporosis, severe hypertension, glaucoma , severe affective disorder and peptic ulceration.

In addition, the following additional exclusion criteria must apply to severe persistent asthmatics with clinical controlled asthma symptoms:

* Changed asthma medication within the 4 weeks prior to screening.
* Has had an asthma exacerbation in the previous month.
* sensitivity or allergy to prednisolone.
* History of tuberculosis, diabetes mellitus, osteoporosis, hypertension, glaucoma, severe affective disorder and peptic ulceration.
* Current use or use within the previous 4 weeks of oral prednisolone or equivalent of greater than 20mg daily.
* Current use of Methotrexate, cyclosporin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-08-02 (Actual); Primary Completion 2011-06-06 (Actual); Study Completion 2011-06-06 (Actual)

PRIMARY OUTCOMES:
Airway pathology endpoints Target Validation endpoints Biomarker endpoints Clinical endpoints | Through 2 weeks of Prednisolone dosing
  biomarkers, vital signs, ECG

SECONDARY OUTCOMES:
Expression of airway and systemic biomarkers. Relationship between changes in target expression and clinical measures of disease activity. Relationship between steady state plasma exposure of prednisolone and pharmacodynamic biomarkers. | Through 2 weeks of prednisolone dosing.
  biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Siddiqui S, Shikotra A, Richardson M, Doran E, Choy D, Bell A, Austin CD, Eastham-Anderson J, Hargadon B, Arron JR, Wardlaw A, Brightling CE, Heaney LG, Bradding P. Airway pathological heterogeneity in asthma: Visualization of disease microclusters using topological data analysis. J Allergy Clin Immunol. 2018 Nov;142(5):1457-1468. doi: 10.1016/j.jaci.2017.12.982. Epub 2018 Mar 14. PMID 29550052
- See also: Results for study RES100769 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/RES100769?search=study&search_terms=RES100769#rs